CLINICAL TRIAL: NCT05263102
Title: Evaluation of the Efficacy and Safety of A High Molecular Weight, Natural Hyaluronic Acid Vaginal Gel in Women With Genitourinary Syndrome of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN Biomedical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAN2014005-CT02
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Menopause Syndrome

STUDY DESIGN:
Intervention Model Description: before and after treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Treatment duration: 8 weeks Twice treatments per week
  Interventions: Device: Vaginal Moisturizing Gel

INTERVENTIONS:
Device: Vaginal Moisturizing Gel — All eligible subjects will received the Vaginal Moisturizing Gel twice per week, total in 8 weeks

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of the vaginal gel with HMW HA in women with genitourinary syndromes due to either menopause or other causes such as the patients after ovarian or breast cancer diagnosis and treatment.

DETAILED DESCRIPTION:
It was recognized that GSM is likely to be underdiagnosed and undertreated9. The North American Menopause Society (NAMS) issued the treatment guideline of GSM in 2014 and encouraged the physicians and nurses to pursue menopausal women to check if they have genitourinary syndrome. GSM is considered a progressive condition in menopausal women, and the primary goal of treatment strategy is symptom relief. Options include lifestyle changes, non-hormonal, and hormonal treatments. Hormonal therapies include both topical and systemic approaches. However, many women reported that substantial concerns about the long-term safety of hormonal products.The patients are aware of the possible relationship between cancer, heart disease, stroke, and estrogen-based treatments10. For considering long-term treatment strategy, estrogen free products of vaginal lubricant or vaginal moisturizer are recommended as first line treatment for those with mild to moderate syndrome.

ELIGIBILITY:
1. Subjects who have the relevant syndromes of vulvovaginal atrophy, and who are

   1. In the status of menopause (≥12 months after the last menstrual cycle); or
   2. FSH > 40 mIU/ml and estradiol level < 20 pg/ml; or
   3. bilateral ovary resection; or
   4. the patients, i.e. breast cancer patients, who completed cancer therapy
2. Subjects have self-identified at least one of mild to moderate or severe symptoms listed below that are the most bothersome to her.

   1. Vaginal dryness
   2. Vaginal and/or vulvar irritation/itching
   3. Dysuria
   4. Vaginal pain associated with sexual activity
   5. Vaginal bleeding associated with sexual activity
3. Subjects are willing to comply with all aspects of the study and have signed informed consent form.

Exclusion Criteria:

1. Subjects have been diagnosed with cervical or vaginal malignant neoplasms
2. Subjects with abnormal undiagnostic genital bleeding
3. Subject with active vaginal infection
4. Subjects with vaginal pH value < 4.5
5. Subjects are under hormone replacement therapy within three months
6. Subjects are under phytoestrogen treatment within two month
7. Subjects use of vaginal douche, lubricant or moisturizer in one week
8. Subjects are hypersensitive to sodium hyaluronate, carrageenan

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who suffer genitourinary syndrome of Menopause
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
pH value change | from baseline to week 8
  The change of the vaginal pH value

SECONDARY OUTCOMES:
The Questionnaire of Genitourinary Syndromes of Menopause | from baseline to week 8
  The change of its severity is used to evaluate symptomatic improvement. The minimum value is 0 and maximum value is 3, where higher scores mean a worse outcome.
Vaginal maturation index (VMI) | from baseline to week 8
  The change of its value is used to evaluate the maturation of the vaginal epithelial cells

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei